CLINICAL TRIAL: NCT05906966
Title: Cognitive, Emotional, Communicative, and Motor Development in Children Born From in Vitro Fertilization of Cryopreserved Oocytes
Brief Title: Cognitive, Emotional, Communicative, and Motor Development in Children Born From IOC
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 1234567
Record Dates: First submitted 2023-03-31; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: ART; Child Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CHILDREN: BORN FROM IN VITRO FERTILIZATION OF CRYOPRESERVED OOCYTES
  Interventions: Other: Phone contact

INTERVENTIONS:
Other: Phone contact — . All mothers of children of born from cryopreserved oocytes will be contacted by phone and administered a questionnaire, to gather additional information about further psychomotor development of children.

SUMMARY:
The study focuses on children born after in vitro fertilization (IVF) of cryopreserved oocytes.

DETAILED DESCRIPTION:
* Evaluate whether the cognitive development of children born by IVF of cryopreserved oocytes is comparable to expected peer development.
* Evaluate whether the emotional development of children born by IVF of cryopreserved oocytes is comparable to expected peer development.
* Evaluate whether the communicative development of children born by IVF of cryopreserved oocytes is comparable to expected peer development.
* Evaluate whether the motor development of children born by IVF of cryopreserved oocytes is comparable to expected peer development

ELIGIBILITY:
Inclusion Criteria:

* Live births from pregnancies resulted from fresh and frozen embryo transfer after fertilization of cryopreserved oocytes are included.

Exclusion Criteria:

* Children born from pregnancies obtained from cryopreserved donated oocytes have been excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Live births from pregnancies resulted from fresh and frozen embryo transfer after fertilization of cryopreserved oocytes are included.
Sampling Method: Probability Sample
Enrollment: 377 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Cognitive development | 18 YEARS
  Evaluation through a newly edited questionnaire according to milestones, set for age, established by CDC guidelines (Zubler et al, 2022). The objective is to compare cognitive development of children born by IVF of cryopreserved oocytes in comparison to expected peer development. Answers will be reported as yes/no according if milestones are achieved or not.
Communicative development | 18 YEARS
  Evaluation through a newly edited questionnaire according to milestones, set for age, established by CDC guidelines (Zubler et al, 2022). The objective is to compare communicative development of children born by IVF of cryopreserved oocytes in comparison to expected peer development. Answers will be reported as yes/no according if milestones are achieved or not.
Motor development | 18 YEARS
  Evaluation through a newly edited questionnaire according to milestones, set for age, established by CDC guidelines (Zubler et al, 2022). The objective is to compare motor development of children born by IVF of cryopreserved oocytes in comparison to expected peer development. Answers will be reported as yes/no according if milestones are achieved or not.
Emotional development | 18 YEARS
  Evaluation through a newly edited questionnaire according to milestones, set for age, established by CDC guidelines (Zubler et al, 2022). The objective is to compare emotional development of children born by IVF of cryopreserved oocytes in comparison to expected peer development. Answers will be reported as yes/no according if milestones are achieved or not.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Emanuele Levi Setti, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy